CLINICAL TRIAL: NCT00095355
Title: Stimulation of Tyrosine Kinase and ERK Signaling Pathways in Huntington's Disease
Brief Title: Effects of Lithium and Divalproex'on Brain-Derived Neurotrophic Factor in Huntington's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050020; 05-N-0020
Record Dates: First submitted 2004-11-02; First posted 2004-11-03 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: Huntington's Disease
Keywords: BDNF; Lithium; Divalproex; Huntington Disease; HD
MeSH Terms: conditions — Huntington Disease | interventions — Lithium; Valproic Acid

INTERVENTIONS:
Drug: Lithium
Drug: Divalproex

SUMMARY:
This study will examine whether lithium carbonate, given alone or with divalproex, increases the amount of brain-derived neurotrophic factor (BDNF) in the spinal fluid of patients with Huntington's disease (HD), a hereditary disorder of the central nervous system. Patients with this fatal degenerative disease have lower amounts of substances in the brain and spinal fluid called trophic or growth factors. One of these factors is BDNF. A possible treatment for HD may be to increase the levels of BDNF. Lithium carbonate, a drug used to treat bipolar disorder, and divalproex, a drug used to treat mood disorders and seizure disorders, have both been shown to increase the amount of BDNF protein in laboratory studies.

Patients 18 to 70 years old with a DNA-confirmed diagnosis of Huntington's disease may be eligible for this study. Candidates are screened with a medical history and physical examination, neurological evaluation, blood and urine tests, and electrocardiogram (EKG).

Participants take lithium carbonate with and without divalproex. They also receive placebo (an inactive substance) for portions of the study. On the first day of the study, patients are given a supply of pills with instructions on how to take them. Blood pressure and pulse are measured, and blood and urine tests may be done. Patients are evaluated with standardized tests and scales for assessment of various aspects of HD.

Patients return to the clinic once a week for follow-up evaluations, including blood and urine tests, physical examinations, disease assessments, and a review of medication side effects. Each week, they receive a new supply of medications and instructions on how to take them. At the end of the sixth week, they finish taking the medications.

During the study, patients undergo three lumbar punctures (spinal taps) - at weeks 2, 4, and 6 - to measure BDNF and various other brain chemicals. For this test, a local anesthetic is given and a needle is inserted in the space between the bones in the lower back where the CSF circulates below the spinal cord. A small amount of fluid is collected through the needle. The procedure generally takes from 5 to 20 minutes.

Patients return to the clinic 2 weeks after completing the study medication for a final evaluation, including a physical examination and blood and urine tests.

DETAILED DESCRIPTION:
Objective: The overall objective of this study is to examine the acute effects of lithium alone and/ or in combination with divalproex on markers of neuroprotective activity in patients with Huntington's disease (HD). It is hypothesized that at safe and tolerable doses these drugs will enhance depleted levels of brain-derived neurotrophic factor (BDNF), a neurotrophin which is necessary for the survival of striatal neurons.

Study population: Patients suffering from Huntington's disease will be study participants.

Design: The acute effects of lithium and divalproex on surrogate measures of neuroprotective activity will be evaluated in up to 24 HD patients. The study, lasting approximately 6 weeks, will be conducted on an outpatient basis.

Outcome measures: In this proof-of-principle study, efficacy in restoring BDNF concentrations will be assessed through cerebrospinal fluid (CSF) measurements. Safety will be monitored by means of frequent clinical evaluations and laboratory test.

ELIGIBILITY:
INCLUSION CRITERIA

1. Subject is between the ages of 18 and 70 (inclusive);
2. Subject will have a diagnosis of HD confirmed by DNA testing [prior to enrollment into the study].
3. Only those subjects will be eligible, who with or without a caregiver, can be assumed to be able to comply with study requirements and to report on their condition by telephone.
4. Subjects with minimental status examination score of greater than and equal to 24.

EXCLUSION CRITERIA

Patients meeting any of the following exclusion criteria during screening or during the study will not be immediately excluded from the study, as appropriate:

1. Patient has a history of any medical condition such as diabetes, cardiac disease, renal impairment, liver disease, pancreatitis and other chronic medical problems that can reasonably be expected to subject the patient to unwarranted risk;
2. Patient has clinically significant laboratory abnormalities that would preclude administration of lithium and divalproex;
3. Patient is taking a prohibited concomitant medication;
4. Patient has not been using an adequate contraceptive method for the last 30 days or unwilling to continue contraception throughout the study, or is not at least one year post menopausal (if female);
5. Patient is pregnant or breastfeeding;
6. Patient has participated in a clinical study with an investigational drug within the last 30 days;
7. Patient has a condition (such as active drug or alcohol abuse) that, in the opinion of the investigators, would interfere with compliance or safety;
8. Patient has known hypersensitivity to lithium or divalproex;
9. Patients inability to swallow tablets or to comply with medication schedule;
10. Patient and / or caregiver are unwilling to sign an informed consent or to comply with protocol requirements;
11. Patient is unwilling to have lumbar puncture.
12. Patient with history of severe depression, or past suicide attemps.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 2004-10; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hedreen JC, Folstein SE. Early loss of neostriatal striosome neurons in Huntington's disease. J Neuropathol Exp Neurol. 1995 Jan;54(1):105-20. doi: 10.1097/00005072-199501000-00013. PMID 7815073
- [Background] A novel gene containing a trinucleotide repeat that is expanded and unstable on Huntington's disease chromosomes. The Huntington's Disease Collaborative Research Group. Cell. 1993 Mar 26;72(6):971-83. doi: 10.1016/0092-8674(93)90585-e. PMID 8458085
- [Background] Bibel M, Barde YA. Neurotrophins: key regulators of cell fate and cell shape in the vertebrate nervous system. Genes Dev. 2000 Dec 1;14(23):2919-37. doi: 10.1101/gad.841400. No abstract available. PMID 11114882